CLINICAL TRIAL: NCT03434587
Title: A Randomized, Open-label Trial to Compare the Functional and Radiological Results of Syndactyly Versus Closed Reduction and Immobilization in Patients With 5th Metacarpal Neck Fracture
Brief Title: Syndactyly Versus Closed Reduction in 5th Metacarpal Neck Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FJD-5MTC-16/01
Record Dates: First submitted 2018-01-26; First posted 2018-02-15 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2017-08

CONDITIONS: Metacarpal Fracture
Keywords: fifth metacarpal neck, fracture, syndactyly, inmobilization, RCT
MeSH Terms: conditions — Fractures, Bone; Syndactyly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Syndactyly (Experimental): Syndactyly
  Interventions: Procedure: Syndactyly
- Reduction and inmobilization (Active Comparator): Closed reduction and splint inmobilization
  Interventions: Procedure: Reduction and inmobilization

INTERVENTIONS:
Procedure: Syndactyly — Syndactyly
  Arms: Syndactyly
Procedure: Reduction and inmobilization — Closed reduction and inmobilization with splint
  Arms: Reduction and inmobilization

SUMMARY:
This study aims to compare the functional results of two different therapeutic approaches in patients that present with a 5th metacarpal neck fracture. Patients will be randomly assigned to be treated with either syndactyly or closed reduction plus inmovilization.

DETAILED DESCRIPTION:
Syndactyly, although limiting the activity of the patient, allows a quick mobilization and recovery, as well as a better management in daily activities compared with immobilization with splint. In addition, follow-up of these fractures is difficult due to poor compliance, since patient profile is young people who give little relevance to their pathology in the hand.

The purpose of our study is to carry out a randomized clinical trial of good methodological quality to assess whether immobilization with syndactyly for 3 weeks does not imply loss of functionality or residual symptoms, avoiding rigidity, postinflammation arthritis or loss of grip strength, demonstrating that early mobilization of fractures of the fifth metacarpal provides clinically satisfactory results compared to prolonged immobilization provided that the volar fracture angle does not exceed 70 ° nor does it produce digital movement disruption.

ELIGIBILITY:
* Inclusion Criteria:
* Men and Women ≥ 18 years old.
* Admitted to the Emergency Department with fracture of 5th metacarpal neck, in acute phase (maximum 72 h of evolution) with a possibility of clinical and radiological follow-up of at least 6 months.
* Willing to participate in the study and give their consent in writing.
* Exclusion Criteria:
* Patients younger than 18 years.
* Patients presenting with more than 72 h of evolution
* Patients with comminuted neck fractures.
* Patients with angulation greater than 70 in the lateral-oblique plane
* Patients with clinical-radiological disruption
* Patients with previous fractures in the metacarpal.
* Patients with open fracture grade II-III Gustilo.
* Patients with bifocal fractures or fractures in another metacarpal-phalanx or carpal bones requiring different treatment.
* Polytraumatized patients requiring further care that prevents them from adjusting to the therapeutic regimen specific to the protocol of isolated metacarpal fractures.
* Patients with congenital anomalies on hand affect
* Patients with a psychic disability (dementia-psychiatric illness or mental disorder) that prevents their collaboration in the follow-up
* Patients with medical or surgical pathologies that at the discretion of the investigator do not allow their participation in the study.
* Patients with inability to understand the nature and purpose of the study and / or to accept written participation in the study.
* Unable to attend the pre-established clinical follow-up.
* Do not wish to participate or give their consent in writing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) score | 9 weeks
  Comparison of DASH score at 9 weeks of emergency care in both treatment groups. Score range is from 0 to 100

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) score | 3 weeks, 1 year
  Comparison of DASH score at 3,6 weeks, 3 months and 1 year of emergency care in both treatment groups.
Time to go back to job and sports | 1 year
  Comparison of the time to incorporation into the work and sports activity between both groups.
Angulation, | 3 weeks, 9 weeks
  Comparison of angulation between both groups
Range of mobility | 3 weeks, 9 weeks
  Comparison of range of mobility between both groups
Grip strength | 3 weeks, 9 weeks
  Comparison of grip strength between both groups
Visual Analogic Scale (VAS) for Pain score | 3 weeks, 9 weeks, 1 year
  Comparison of VAS score
Complication rate | 1 year
  Frequency of complications
Patient satisfaction (Modified Cooney Scale) | 1 year
  Satisfaction with the assigned treatment and its result between groups, measured by the modified cooney scale that ranges from 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Pajares, MD, Principal Investigator — IIS-FJD
Locations (1):
- Fundacion Jimenez Diaz, Madrid, Spain